CLINICAL TRIAL: NCT05564676
Title: Effects of Supplementation With Flaxseed Oil and Pomegranate Extract on Inflammation Markers, Lipid Profile and Nutritional Status of Individuals on Hemodialysis: a Randomized, Placebo-controlled, Triple-blind Clinical Trial
Brief Title: Flaxseed Oil and Pomegranate Extract on Inflammation, Lipid Profile and Nutritional Status of Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Catarina Federal University (Other)
Responsible Party: Principal Investigator, Aline Miroski de Abreu, Principal investigator, Santa Catarina Federal University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UFSC
Record Dates: First submitted 2022-09-04; First posted 2022-10-03 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Chronic Kidney Diseases; Dialysis; Complications; Inflammation; Lipid Metabolism Disorders
Keywords: Chronic kidney disease; hemodialysis; inflammation; dyslipidemia; flaxseed; pomagranate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation; Lipid Metabolism Disorders; Dyslipidemias | interventions — Linseed Oil; Sunflower Oil; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- flaxseed oil and pomegranate extract (Experimental): 2g daily of flaxseed oil plus 1.2g daily pomegranate dry extract
  Interventions: Dietary Supplement: flaxseed oil and pomegranate dry extract
- sunflower oil and microcrystalline cellulose (Placebo Comparator): 2g daily of sunflower oil plus 1.2g daily microcrystalline cellulose
  Interventions: Dietary Supplement: sunflower oil and microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: flaxseed oil and pomegranate dry extract — The flaxseed oil were yellow capsules with 1.0 g each and the pomegranate dry extract capsules were green with 0.6 g each.
  Arms: flaxseed oil and pomegranate extract
Dietary Supplement: sunflower oil and microcrystalline cellulose — The sunflower oil were yellow capsules with 1.0 g each and the microcrystalline cellulose capsules were green with 0.6 g each.
  Arms: sunflower oil and microcrystalline cellulose

SUMMARY:
Nutritional and metabolic alterations in patients with chronic kidney disease (CKD) such as inflammation, oxidative stress, dyslipidemia, and poor nutritional status which associate with poor clinical outcome can potentially be targeted and ameliorated by interventions using nutritional supplements. The investigators evaluated the effects of 8 weeks of oral supplementation with flaxseed oil and pomegranate dry extract on markers of inflammation, lipid profile and nutritional status of individuals undergoing hemodialysis (HD).

The goal of this randomized, placebo-controlled, double-blind clinical trial is to evaluate the effects of 8 weeks of oral supplementation with flaxseed oil and pomegranate dry extract on markers of inflammation, lipid profile and nutritional status of individuals undergoing hemodialysis (HD).

Participants will be randomly assigned, in a 1:1 ratio, to supplementation group to receive twice a day 1 capsule of 1.000 mg of flaxseed oil plus 1 capsule of 600mg of pomegranate dry extract; or to placebo group, to receive twice a day 1 capsule of 1.000 mg of sunflower oil plus 1 capsule of 600mg of microcrystalline celulose.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 19 years; have a diagnosis of CKD;
* perform HD three times a week for a period of ≥ three months;
* acceptance of participation.

Exclusion Criteria:

* history of allergy to flaxseed or pomegranate;
* infection or hospitalization in the beginning or during the course of the study;
* HIV seropositivity and active malignancy;
* pregnancy or breastfeeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
interleukin 2 | Change from Baseline and at 8 weeks (end of study)
interleukin 4 | Change from Baseline and at 8 weeks (end of study)
interleukin 6 | Change from Baseline and at 8 weeks (end of study)
interleukin 10 | Change from Baseline and at 8 weeks (end of study)
tumor necrosis factor alpha | Change from Baseline and at 8 weeks (end of study)
interferon-gamma | Change from Baseline and at 8 weeks (end of study)
C-reactive protein | Change from Baseline and at 8 weeks (end of study)

SECONDARY OUTCOMES:
total cholesterol | Change from Baseline and at 8 weeks (end of study)
high-density lipoprotein | Change from Baseline and at 8 weeks (end of study)
low-density lipoprotein | Change from Baseline and at 8 weeks (end of study)
triglycerides | Change from Baseline and at 8 weeks (end of study)

OTHER OUTCOMES:
weight | Change from Baseline and at 8 weeks (end of study)
height | Change from Baseline and at 8 weeks (end of study)
handgrip strength | Change from Baseline and at 8 weeks (end of study)
waist circumference | Change from Baseline and at 8 weeks (end of study)
calf circumference | Change from Baseline and at 8 weeks (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Aline M de Abreu, MSc, Principal Investigator — UFSC
Locations (1):
- Federal University of Santa Catarina, Florianópolis, Santa Catarina, Brazil